CLINICAL TRIAL: NCT05918900
Title: Descriptive and Comparative Analyses of Malnutrition Screening in Internal Medicine
Brief Title: Analyses of Malnutrition Screening in Internal Medicine
Acronym: AMASIN
Status: Completed | Type: Observational
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Other Study IDs: BB 073/23
Record Dates: First submitted 2023-06-15; First posted 2023-06-26 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Malnutrition
Keywords: Malnutrition risk; Screening; Internal medicine; Nutritional Risk Screening 2002; Gastroenterology; Nephrology; Endocrinology; Rheumatology
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to study the presence and consequences of malnutrition risk in hospitalized internal medicine patients.

The main questions it aims to answer are:

1. How many patients are at risk of malnutrition at admission?
2. Is there a link between an existing malnutrition risk and nutrition therapy that the patients receive?
3. Is there a link between an existing malnutrition risk and clinical outcome (e.g. length of hospital stay, mortality, need for rehospitalization)?

Participants will be screened for malnutrition risk at admission using a validated questionnaire (Nutritional Risk Screening 2002). All relevant data regarding hospital stay will be obtained from the clinical information system after discharge.

DETAILED DESCRIPTION:
Malnutrition is associated with adverse clinical outcome in hospitalized patients. Therefore, systematic screening for malnutrition risk at admission is recommended by almost all medical expert societies to identify patients who will benefit from nutritional therapy.

Although clinical and economic benefit of systematic malnutrition screening have been shown in various settings and for different patient groups, such screening is still not mandatory in most countries. In part, establishment of malnutrition screening is hampered by discrepant findings on the prevalence of malnutrition risk and the lack of evidence on a local level.

Hence, in this observational study the investigators examine the results of systematic malnutrition screening in internal medicine patients admitted to a university hospital in Northeast Germany. In particular, the investigators aim to determine the prevalence of malnutrition risk at hospital admission, the association between malnutrition risk and nutrition therapy as well as clinical outcome in different disciplines of internal medicine.

For this purpose, all patients undergo screening for malnutrition risk at admission using a validated instrument (Nutritional Risk Screening 2002). All relevant data regarding the patients' hospital stay will be obtained from the clinical information system after discharge.

ELIGIBILITY:
Inclusion Criteria:

* hospital admission for gastrointestinal, endocrine, rheumatic, or nephrological condition
* provision of informed consent

Exclusion Criteria:

* inability to provide consent
* unfeasibility to perform malnutrition screening within 48h after admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited at University Medicine Greifswald (Northeast Germany). Internal medicine patients with any gastrointestinal, endocrine, rheumatic, or nephrological disease admitted to the hospital will be identified in the respective wards and will be approached for study inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 323 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2023-09-22 (Actual)

PRIMARY OUTCOMES:
Overall presence of malnutrition risk | Baseline
  Prevalence of malnutrition risk, i.e. Nutritional Risk Screening 2002 (NRS-2002) score >= 3 points, in all internal medicine patients at hospital admission. NRS-2002 score ranges from 0 to 7, with higher values indicating greater nutritional risk.

SECONDARY OUTCOMES:
Presence of malnutrition risk in gastroenterology | Baseline
  Prevalence of malnutrition risk, i.e. Nutritional Risk Screening 2002 (NRS-2002) score >= 3 points, in patients with gastrointestinal disease at hospital admission. NRS-2002 score ranges from 0 to 7, with higher values indicating greater nutritional risk.
Presence of malnutrition risk in endocrinology | Baseline
  Prevalence of malnutrition risk, i.e. Nutritional Risk Screening 2002 (NRS-2002) score >= 3 points, in patients with endocrine disease at hospital admission. NRS-2002 score ranges from 0 to 7, with higher values indicating greater nutritional risk.
Presence of malnutrition risk in rheumatology | Baseline
  Prevalence of malnutrition risk, i.e. Nutritional Risk Screening 2002 (NRS-2002) score >= 3 points, in patients with rheumatic disease at hospital admission. NRS-2002 score ranges from 0 to 7, with higher values indicating greater nutritional risk.
Presence of malnutrition risk in nephrology | Baseline
  Prevalence of malnutrition risk, i.e. Nutritional Risk Screening 2002 (NRS-2002) score >= 3 points, in patients with nephrological disease at hospital admission. NRS-2002 score ranges from 0 to 7, with higher values indicating greater nutritional risk.
Relation of malnutrition risk to nutritional consultation | Baseline
  Association between malnutrition risk, i.e. Nutritional Risk Screening 2002 (NRS-2002) score >= 3 points, and number of nutritional consultations. NRS-2002 score ranges from 0 to 7, with higher values indicating greater nutritional risk.
Relation of malnutrition risk to nutritional diagnosis | Baseline
  Association between malnutrition risk, i.e. Nutritional Risk Screening 2002 (NRS-2002) score >= 3 points, and nutritional diagnosis resulting from nutritional assessment by an expert dietitian. NRS-2002 score ranges from 0 to 7, with higher values indicating greater nutritional risk.
Relation of malnutrition risk to intensive care treatment | Baseline
  Association between malnutrition risk, i.e. Nutritional Risk Screening 2002 (NRS-2002) score >= 3 points, and admission to an intensive care unit. NRS-2002 score ranges from 0 to 7, with higher values indicating greater nutritional risk.
Relation of malnutrition risk to intermediate care treatment | Baseline
  Association between malnutrition risk, i.e. Nutritional Risk Screening 2002 (NRS-2002) score >= 3 points, and admission to an intermediate care unit. NRS-2002 score ranges from 0 to 7, with higher values indicating greater nutritional risk.
Relation of malnutrition risk to mortality | Baseline
  Association between malnutrition risk, i.e. Nutritional Risk Screening 2002 (NRS-2002) score >= 3 points, and in-hospital mortality. NRS-2002 score ranges from 0 to 7, with higher values indicating greater nutritional risk.
Relation of malnutrition risk to length of hospital stay | Baseline
  Association between malnutrition risk, i.e. Nutritional Risk Screening 2002 (NRS-2002) score >= 3 points, and length of hospital stay measured in days. NRS-2002 score ranges from 0 to 7, with higher values indicating greater nutritional risk.
Relation of malnutrition risk and 30-day readmission | Baseline
  Association between malnutrition risk, i.e. Nutritional Risk Screening 2002 (NRS-2002) score >= 3 points, and unplanned hospital readmission within 30 days after discharge. NRS-2002 score ranges from 0 to 7, with higher values indicating greater nutritional risk.
Relation of malnutrition risk and 90-day readmission | Baseline
  Association between malnutrition risk, i.e. Nutritional Risk Screening 2002 (NRS-2002) score >= 3 points, and unplanned hospital readmission within 90 days after discharge. NRS-2002 score ranges from 0 to 7, with higher values indicating greater nutritional risk.

CONTACTS AND LOCATIONS:
Overall Officials: Ali A Aghdassi, Professor, Principal Investigator — University Medicine Greifswald
Locations (1):
- University Medicine Greifswald, Greifswald, Germany